CLINICAL TRIAL: NCT00077857
Title: A Randomized, Open-label Study of the Effect of Different Dosing Regimens of Xeloda® in Combination With Taxotere® on Disease Progression in Patients With Locally Advanced and/or Metastatic Breast Cancer
Brief Title: A Study to Assess Capecitabine (Xeloda®) in Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO16853; NCT00083200 (obsolete NCT alias)
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Results first posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel

ARMS (2):
- 1250 mg/m^2 capecitabine + docetaxel (Experimental): 1250 mg/m^2 capecitabine (Xeloda®) orally twice a day on days 1 to 14 of each 3 week cycle, in combination with docetaxel (Taxotere®) 75 mg/m^2 intravenous on day 1 of each 3 week cycle.
  Interventions: Drug: capecitabine (Xeloda®); Drug: docetaxel (Taxotere®)
- 825 mg/m^2 capecitabine + docetaxel (Experimental): 825 mg/m^2 capecitabine orally twice a day on days 1 to 14 of each 3 week cycle, in combination with docetaxel 75 mg/m^2 intravenous on day 1 of each 3 week cycle.
  Interventions: Drug: capecitabine (Xeloda®); Drug: docetaxel (Taxotere®)

INTERVENTIONS:
Drug: capecitabine (Xeloda®) — 825 mg/m^2 or 1250 mg/m2 orally twice a day on days 1 to 14 of each 3 week cycle.
  Other Names: Xeloda®
Drug: docetaxel (Taxotere®) — 75 mg/m^2 intravenous on day 1 of each 3 week cycle
  Other Names: Taxotere®

SUMMARY:
This 2 arm study compared the efficacy and safety of label dose of capecitabine (Xeloda®) to that of a lower dose of Xeloda® plus docetaxel (Taxotere®) in patients with locally advanced or metastatic breast cancer after failure of chemotherapy with an anthracycline. Patients were randomized to receive either 1250 mg/m^2 or 825 mg/m^2 orally twice a day (po bid) on days 1-14 of each 3 week cycle, in combination with Taxotere® 75 mg/m2 intravenous (iv) on day 1 of each 3 week cycle. The anticipated time on study treatment was until disease progression and the target sample size was 440 individuals.

ELIGIBILITY:
Inclusion Criteria:

* women >=18 years of age;
* >=1 target lesion;
* locally advanced or metastatic breast cancer;
* demonstrated resistance to anthracycline;
* >=2 regimens of chemotherapy for advanced/metastatic disease.

Exclusion Criteria:

* previous treatment with Xeloda, continuous 5-fluorouracil infusion, or other oral fluoropyrimidines;
* previous treatment with paclitaxel or docetaxel for advanced/metastatic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2003-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (83):
- United States (42):
  - Birmingham, Alabama
  - Hoover, Alabama
  - Tucson, Arizona
  - Berkeley, California
  - Poway, California
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Miami Shores, Florida
  - Port Saint Lucie, Florida
  - Tamarac, Florida
  - Skokie, Illinois
  - Urbana, Illinois
  - Beech Grove, Indiana
  - Des Moines, Iowa
  - Overland Park, Kansas
  - Houma, Louisiana
  - Baltimore, Maryland
  - Frederick, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Jefferson City, Missouri
  - Saint Joseph, Missouri
  - Paramus, New Jersey
  - Summit, New Jersey
  - Williamsville, New York
  - Canton, Ohio
  - Mayfield Heights, Ohio
  - Allentown, Pennsylvania
  - Kingston, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Collierville, Tennessee
  - Knoxville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Colchester, Vermont
  - Abingdon, Virginia
  - Walla Walla, Washington
- Bosnia and Herzegovina (3):
  - Mostar
  - Sarajevo
  - Tuzla
- China (6):
  - Beijing
  - Bengbu
  - Dalian
  - Hangzhou
  - Shanghai
  - Tianjin
- Czechia (3):
  - Pardubice
  - Prague
  - Tábor
- India (12):
  - Ahmedabad
  - Bangalore
  - Hyderabad
  - Jaipur
  - Kochi
  - Kolkata
  - Ludhiana
  - Manipal
  - Mumbai
  - New Delhi
  - Trivandrum
  - Vellore
- Poland (2):
  - Poznan
  - Wroclaw
- Russia (9):
  - Chelyabinsk
  - Ivanovo
  - Kazan'
  - Moscow
  - Omsk
  - Ryazan
  - Saint Petersburg
  - Samara
  - Yaroslavl
- South Africa (3):
  - Bloemfontein
  - Durban
  - Polokwane
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Started | 235 | 235
Received Study Drug | 231 | 234
Safety Population: Actual Dose Received | 217 (14 patients in the 1250 dose arm received a lower dose and were included in the 825 arm for Safety.) | 248
Completed | 34 | 31
Not Completed | 201 | 204
Not completed — Adverse Event | 30 | 32
Not completed — Death | 7 | 3
Not completed — Insufficient therapeutic response | 112 | 128
Not completed — Violation of selection criteria at entry | 3 | 1
Not completed — Other protocol violation | 0 | 1
Not completed — Refused treatment | 29 | 21
Not completed — Failure to return | 5 | 5
Not completed — Other | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel | Total
Number analyzed (Participants) | 235 | 235 | 470
Age Continuous [Mean (Full Range); unit: years] | 50.9 [22 to 75] | 50.6 [28 to 75] | 50.75 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235 | 235 | 470
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression of Disease or Death
Description: Progression Free Survival was defined as the time from the date of randomization to the day of documented disease progression or death due to any cause.
Time Frame: Event driven (after 350 events). Median observation time was approximately 16 months.
Population: Per protocol population included all participants who received at least one dose of study and who did not have any major protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 230 | 229
Months | 7.9 [6.9 to 8.5] | 5.8 [4.9 to 7.1]

2. Secondary Outcome: Percentage of Participants With Best Overall Response Being Complete Response (CR) or Partial Response (PR)
Description: According to Response Evaluation Criteria in Solid Tumors (RECIST) criteria: CR is defined as the disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the nadir sum LD.
Time Frame: Until Progressive Disease (PD) or end of primary study treatment (up to 16 cycles) plus 28 days.
Population: Intent to treat population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 235 | 235
Percentage of participants | 45.1 [38.6 to 51.7] | 37.4 [31.2 to 44.0]

3. Secondary Outcome: Time to Overall Response
Description: For patients with Best Overall Response being Complete Response (CR) or Partial Response (PR), time to response was measured as the time from randomization to the first time when the measurement criteria for CR or PR were met. The percentage of participants with overall response within the given time ranges in each of the categories: Weeks 1-6, 7-12, 13-18, 19-24, 25-30, 31-36, and 43-48 are reported.
Time Frame: Until PD or end of primary study treatment (up to 16 cycles) plus 28 days.
Population: Intent to treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 235 | 235
Percentage of participants
  Week 1-6 | 25 | 30
  Week 7-12 | 48 | 30
  Week 13-18 | 20 | 17
  Week 19-24 | 7 | 7
  Week 25-30 | 3 | 1
  Week 31-36 | 3 | 2
  Week 43-48 | 0 | 1

4. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response was measured from the time that measurement criteria were first met for Complete Response or Partial Response until the first date that progressive disease or death was documented.
Time Frame: Until PD or death. Median duration of response was approximately 7 months.
Population: Intent to treat population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 235 | 235
Months | 6.9 [6.1 to 8.6] | 6.9 [5.8 to 9.0]

5. Secondary Outcome: Time to Treatment Failure
Description: The time to treatment failure was the time from the date of randomization to the first occurrence of any of the following events:
  * adverse events
  * insufficient therapeutic response (disease progression)
  * death
  * failure to return
  * refusing treatment/being unwilling to cooperate
  * withdrawing consent.
Time Frame: Until premature withdrawal or end of primary study treatment (up to 16 cycles).
Population: Safety Population included all randomized participants who received study drug. Note: 14 patients randomized to 1250 mg/m^2 actual received an initial dose that ranged from 480 to 984 mg/m^2 so are included in the 825 mg/m^2 arm for safety.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 217 | 248
Months | 5.1 [4.2 to 5.8] | 4.6 [4.1 to 5.3]

6. Secondary Outcome: Overall Survival
Description: Overall Survival was measured as the time from the date of randomization to the date of death.
Time Frame: Throughout the study. Median observation time was approximately 16 months.
Population: Intent to treat population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 235 | 235
Months | 16.4 [13.6 to 21.8] | 15.1 [12.9 to 17.7]

7. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
  A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is Life-Threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
  Additional information about Adverse Events can be found in the Adverse Event Section.
Time Frame: First study drug intake until last study drug intake plus 28 days
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Number analyzed (Participants) | 217 | 248
Participants
  Adverse Events | 206 | 234
  Serious Adverse Events | 41 | 53

ADVERSE EVENTS:
Description: Safety Population included all randomized participants who received study drug. Note: 14 patients randomized to the 1250 mg/m^2 arm actual received an initial dose that ranged from 480 to 984 mg/m^2 so were included in the 825 mg/m^2 arm for safety.
Arm/Group | 1250 mg/m^2 Capecitabine + Docetaxel | 825 mg/m^2 Capecitabine + Docetaxel
Serious Adverse Events (participants affected / at risk) | 41/217 | 53/248
Other Adverse Events (participants affected / at risk) | 192/217 | 223/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1250 mg/m^2 Capecitabine + Docetaxel (N=217) | 825 mg/m^2 Capecitabine + Docetaxel (N=248)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 14
Neutropenia (Blood and lymphatic system disorders) | 6 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Stomatitis all (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 3
Disease progression (General disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 2
Injection site reaction (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Chest wall abscess (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1250 mg/m^2 Capecitabine + Docetaxel (N=217) | 825 mg/m^2 Capecitabine + Docetaxel (N=248)
Stomatitis all (Gastrointestinal disorders) | 87 | 88
Diarrhoea (Gastrointestinal disorders) | 73 | 81
Nausea (Gastrointestinal disorders) | 45 | 58
Vomiting (Gastrointestinal disorders) | 33 | 45
Constipation (Gastrointestinal disorders) | 17 | 17
Abdominal pain (Gastrointestinal disorders) | 14 | 9
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 102 | 104
Alopecia (Skin and subcutaneous tissue disorders) | 74 | 82
Nail disorder (Skin and subcutaneous tissue disorders) | 26 | 38
Rash (Skin and subcutaneous tissue disorders) | 14 | 13
Fatigue (General disorders) | 58 | 50
Pyrexia (General disorders) | 35 | 27
Asthenia (General disorders) | 26 | 34
Oedema peripheral (General disorders) | 18 | 26
Neutropenia (Blood and lymphatic system disorders) | 77 | 70
Leukopenia (Blood and lymphatic system disorders) | 21 | 17
Anaemia (Blood and lymphatic system disorders) | 13 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Decreased appetite (Metabolism and nutrition disorders) | 30 | 36
Blood bilirubin increased (Investigations) | 18 | 15
Aspartate aminotransferase increased (Investigations) | 11 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 31
Headache (Nervous system disorders) | 14 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.